CLINICAL TRIAL: NCT01208818
Title: Treatment of Renal Failure Due to Myeloma Cast Nephropathy: Comparison of Two Different Chemotherapy Regimens and Evaluation of Optimized Removal of Monoclonal Immunoglobulin Light Chains Using a High Permeability Hemodialysis Membrane.
Brief Title: Studies in Patients With Multiple Myeloma and Renal Failure Due to Myeloma Cast Nephropathy
Acronym: MYRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P081226
Record Dates: First submitted 2010-09-23; First posted 2010-09-24 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Chronic Renal Failure With Uremic Nephropathy
MeSH Terms: interventions — Cyclophosphamide; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- BD (Active Comparator)
  Interventions: Drug: Bortezomib +Dexamethasone regimen
- C-BD (Experimental)
  Interventions: Drug: Cyclophosphamide + Bortezomib + Dexamethasone regimen
- HCO (Experimental)
  Interventions: Drug: Bortezomib +Dexamethasone regimen; Device: HCO group
- Control HD (Active Comparator)
  Interventions: Drug: Bortezomib +Dexamethasone regimen; Device: conventional high-flux dialyzer

INTERVENTIONS:
Drug: Cyclophosphamide + Bortezomib + Dexamethasone regimen — Dosing regimen (21 day-cycle):
  * Bortezomib 1.3 mg/m2 I.V. on days 1, 4, 8, and 11. An interval of at least 72 hours between each administration of bortezomib is required.
  * Dexamethasone 20 mg on days 1, 2, 4, 5, 8, 9, 11 and 12.
  * Cyclophosphamide 900 mg/m2 on day 1, through a short I.V. infusion The regimen is given for 3 cycles in the absence of serious side-effect.
  Arms: C-BD
Drug: Bortezomib +Dexamethasone regimen — Dosing regimen (21 day-cycle):
  * Bortezomib 1.3 mg/m2 I.V. on days 1, 4, 8, and 11. An interval of at least 72 hours between each administration of bortezomib is required.
  * Dexamethasone 20 mg on days 1, 2, 4, 5, 8, 9, 11 and 12. The regimen is given for 3 cycles in the absence of serious side-effect.
  Arms: BD; Control HD; HCO
Device: HCO group — TheraliteTM dialyzer of 2.1 m2 in surface
  Arms: HCO
Device: conventional high-flux dialyzer — conventional high-flux dialyzer; polyacrylonitrile, polysulfone, or PMMA dialysers, with an ultrafiltration coefficient > 14 ml/min and ≥ 1.8 m2 in surface, are recommended.
  Arms: Control HD

SUMMARY:
MYRE is a phase III multicentric controlled national clinical trial conducted in patients with multiple myeloma and renal failure related to myeloma cast nephropathy (MCN). Its aims are to assess (1) the efficacy of bortezomib plus dexamethasone (BD), compared with cyclophosphamide, plus bortezomib and dexamethasone (C-BD) in patients with inaugural MCN not requiring hemodialysis; and (2) in patients with inaugural severe renal failure secondary to biopsy-proven MCN and requiring hemodialysis that of an intensive hemodialysis regimen using either a dialyser with very high permeability to proteins (TheraliteTM) or a conventional high-flux dialyser, while receiving chemotherapy with BD.

DETAILED DESCRIPTION:
MYRE is a phase III multicentric controlled national clinical trial conducted in patients with multiple myeloma and renal failure related to myeloma cast nephropathy (MCN). Its aims are to assess (1) the efficacy of bortezomib plus dexamethasone (BD), compared with cyclophosphamide, plus bortezomib and dexamethasone (C-BD) in patients with inaugural MCN not requiring hemodialysis; and (2) in patients with inaugural severe renal failure secondary to biopsy-proven MCN and requiring hemodialysis that of an intensive hemodialysis regimen using either a dialyser with very high permeability to proteins (TheraliteTM) or a conventional high-flux dialyser, while receiving chemotherapy with BD.

Study hypotheses are: (1) in patients not requiring dialysis, based on renal response after 3 cycles as the main endpoint, to show a benefit of 30% in absolute rate from an expected 30% response rate in the control arm; and (2) in patients requiring hemodialysis, using the prevalence of patients free of dialysis after 3 cycles as the main endpoint, to show a benefit of at least 20% from an assumed rate of 50% in the control arm. A total sample size of 284 patients was computed to be enrolled (type I and II error rates at 5 and 20%, respectively).

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years old
* Serum creatinine > 170µmol/l and/or DFG < 40 ml/min/1.73 m2
* Myeloma cast nephropathy (MCN)
* Multiple myeloma
* Informed consent
* neutrophils >= 1 Giga/L and platelets >= 70 Giga/L

Exclusion Criteria:

* Amylosis
* Chronic renal Failure with eDFG < 30 ml/min/1.73 m2, unrelated to myeloma
* Peripheral neuropathy
* Contraindications to either corticosteroids or Bortezomib
* Patient refusal
* Known HIV infection
* Concomitant severe disease including neoplasias (except basocellular carcinoma)
* Liver failure, cytolysis, and/or cholestasis
* Fertile women who refuse or cannot use effective contraception; Women pregnant or nursing; Women with positive test pregnancy (test before treatment initiation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Estimated)
Dates: Start 2011-06; Primary Completion 2015-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of renal response (if dialysis not mandatory at baseline: strata 1); Prevalence of patients free of dialysis (if dialysis required at baseline; strata 2) | 3 months after randomization
  * renal response is defined by creatinine≤ 170 µmol/l and/or DFG (modified MDRD) ≥ 40 ml/min/1.73m2
  * the absence of any dialysis requirement will be defined by an eDFG > 15 ml/min/1.73 m2, 15 days after the last hemodialysis session

SECONDARY OUTCOMES:
Improvement in renal function | after 1 cycle of chemotherapy, at the end of chemotherapy, at 6 months and 1 year
  * DFG (modified MDRD)
  * hemodialysis requirement
Hematological response | after 1 and 3 courses, at the end of chemotherapy and at 1 year
  Partial Response (PR) Very Good Partial Response (VGPR) Complete Response (CR)
Progression free survival (PFS) | 4 years
  Time to progression, relapse or death from randomization
Time to treatment Failure (TTF) | 4 years
  Time from randomization to progression, relapse, non scheduled hematological treatment or death
Overall survival (OS) | 4 years
  Time to death from randomization

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Fermand, MD, Principal Investigator — Hôpital saint Louis, Paris, France; Franck Bridoux, MD, PhD, Study Director — CHU Poitiers
Locations (1):
- Hôpital Saint Louis, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bridoux F, Carron PL, Pegourie B, Alamartine E, Augeul-Meunier K, Karras A, Joly B, Peraldi MN, Arnulf B, Vigneau C, Lamy T, Wynckel A, Kolb B, Royer B, Rabot N, Benboubker L, Combe C, Jaccard A, Moulin B, Knebelmann B, Chevret S, Fermand JP; MYRE Study Group. Effect of High-Cutoff Hemodialysis vs Conventional Hemodialysis on Hemodialysis Independence Among Patients With Myeloma Cast Nephropathy: A Randomized Clinical Trial. JAMA. 2017 Dec 5;318(21):2099-2110. doi: 10.1001/jama.2017.17924. PMID 29209721